CLINICAL TRIAL: NCT02608827
Title: Sympathetic and Blood Pressure Responses to Aerobic Exercise and Guided Respiration in Hypertensives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Tatiana Goveia de Araújo, Post graduate, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAPESP 2010/11413-6
Record Dates: First submitted 2015-10-07; First posted 2015-11-20 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension
Keywords: Hypertension; slow breathing; sympathetic nerve activity
MeSH Terms: conditions — Hypertension; Hypoventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Slow breathing group (GRL) (Active Comparator): After randomization and have done aerobic exercise, patients allocated in this arm of the study, using the device-guided breathing - Slow breathing group (GRL), for 15 minutes during the experimental session.
  Interventions: Device: Resperate®-InterCure Ltda
- Music group (GC) (Placebo Comparator): After randomization and have done aerobic exercise, patients allocated in this study arm will hear slow music - Music group (GC), for 15 minutes during the experimental session.
  Interventions: Other: Music group (GC)

INTERVENTIONS:
Device: Resperate®-InterCure Ltda — The device-guided breathing - Resperate®-InterCure Ltda, uses sound to guide and therefore reduce the respiration rate in individuals.
  Arms: Slow breathing group (GRL)
Other: Music group (GC) — The patients in this arm will hear slow music - Music group (GC).
  Arms: Music group (GC)

SUMMARY:
Hypertension is serious health problem in Brazil and affects almost 30%of adult population. It is known that there are pharmacologic and nonpharmacologic strategies for treating hypertension. Aerobic exercise and slow breathing are nonpharmacologic methods that reduce blood pressure in an isolated form, but its combinations has never been studied. The aim of this study is to evaluate the association of both strategies and also the mechanisms involved in blood pressure reduction using slow breathing, in stages 1 and 2 hypertensives.

DETAILED DESCRIPTION:
The combination of drugs and no medication for hypertension treatment has been widely recommended, with emphasis on aerobic exercises (EXE), relaxation exercises, and the use of equipment designed to decrease the respiratory rate called Resperate®. This intervention has demonstrated a hypotensive effect in pressure measurements in clinical blood pressure and ambulatory blood pressure monitoring (ABPM) and home blood pressure monitoring (HBPM). It is unknown; however, if slow breathing (GRL) associated with other intervention, such as EXE, for example, may potentiate the blood pressure (BP) reduction. The aim of this study will be evaluate the acute responses of muscle sympathetic nerve activity (MSNA) and BP, in association of the slow breathing versus control (listening to calm music) and the 24 hour blood pressure response after the association of EXE and GRL. Twenty hypertensives will be evaluated between 18 to 60 years old, mens and woman, sedentary, non-obese, without target organs damage and associated comorbidities, after 4 weeks of placebo use (washout period). Participants will be randomly divided into 2 groups (GRL and GC) and both perform EXE on a cycle ergometer. Volunteers will make a ABPM before and after the experimental session. In this session will be recorded for 10 minutes, prior to the physical exercise, the systolic blood pressure (SBP), diastolic blood pressure (DBP), respiratory rate (RR) and heart rate (HR), after that, It will be held microneurography to register also the MSNA for 10 minutes, then they will perform either GRL or listened to music for 15 minutes. Variables will be measures for more 10 minutes. After finishing the session, volunteers will put the ABPM and will go away.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 60 years, of both sexes not obese (BMI <30 kg / m2);
* Sedentary not to perform physical exercise for at least three months;
* Hypertensive without target organ damage or untreated stage I and stage II (SBP 140-179 mmHg and DBP 90-109 mmHg) after four weeks with the use of placebo and without comorbidities; What would agree to participate in the study by signing the Instrument of Consent;

Exclusion Criteria:

* Patients who presented blood pressure greater than 180/100 mmHg at any rate during the home monitoring of blood pressure and they needed treatment with active drug;
* White-coat hypertension, or persistently elevated BP measurements (≥ 140/90 mmHg) in the office and BP means be considered normal in HBPM or ABPM.
* Masked Hypertension, or high blood pressure office <140/90 mmHg, and 24-hour ABPM with daytime BP> 130/85 mmHg;
* Patients with a history of alcoholism, drug abuse or mental disorders that could invalidate the consent, or limit the patient's ability to comply with the rules of the Protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure reduction | A session (1 day), after the placebo period of 30 days.
  The reduction in blood pressure in mmHg immediately after after a single session of the association of aerobic exercise and guided slow breathing and during 24 hours blood pressure monitoring (ABPM).

SECONDARY OUTCOMES:
Autonomic regulation | A session (1 day), after the placebo period of 30 days.
  The sympathetic nerve activity will be measured by microneurography technique (burst/min), after a single session of bike aerobic exercise and slow breathing with a guided device.

IPD SHARING:
Plan to Share IPD: Undecided